CLINICAL TRIAL: NCT00002145
Title: Phase III Multicenter, Open-Label, Randomized Trial of Induction Versus Induction Plus Maintenance Foscarnet ( Foscavir ) Therapy for Gastrointestinal CMV Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020I; 93-FOS-29
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections; Gastrointestinal Diseases
Keywords: Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Gastrointestinal Diseases; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
PRIMARY: To compare the frequency of and time to relapse of Cytomegalovirus (CMV) gastrointestinal disease following foscarnet induction therapy only versus induction plus maintenance therapy.

SECONDARY: To determine frequency of and time to recurrence of gastrointestinal symptoms, response rate of pathological lesions, and incidence of nongastrointestinal CMV disease in this patient population.

DETAILED DESCRIPTION:
Patients receive intravenous foscarnet either as induction only for 4 weeks or as induction for 4 weeks followed by maintenance for 22 weeks. All patients are followed for 26 weeks or until relapse.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS.
* CMV GI disease.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Non-GI CMV disease.
* Ulcerative colitis, inflammatory bowel disease, or other condition that may interfere with study results.
* Other GI pathogens.

Concurrent Medication:

Excluded:

* Drugs that may interact with foscarnet.
* Systemic acyclovir, ganciclovir, or acyclovir prodrug.
* Drugs known to affect renal function.

Prior Medication:

Excluded:

* Prior foscarnet in extremis.
* Investigational agents other than 3TC or d4T within 7 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - East Bay AIDS Ctr, Berkeley, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Dr Robert Bresalier / Henry Ford Hosp, Detroit, Michigan
  - Dr Douglas Dieterich, New York, New York
  - Dept of Veterans Affairs, Northport, New York
  - Ohio State Univ Hosp, Columbus, Ohio
  - Comprehensive Care Ctr, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Med College of Virginia, Richmond, Virginia

REFERENCES:
- [Background] Dieterich DT, Poles MA, Lew EA, Martin-Munley S, Johnson J, Nix D, Faust MJ. Treatment of gastrointestinal cytomegalovirus infection with twice-daily foscarnet: a pilot study of safety, efficacy, and pharmacokinetics in patients with AIDS. Antimicrob Agents Chemother. 1997 Jun;41(6):1226-30. doi: 10.1128/AAC.41.6.1226. PMID 9174175